CLINICAL TRIAL: NCT05882435
Title: Intelligence for the Interpretation of Bone Standard X-rays Prescribed by the Emergency Department
Brief Title: Use of Augmented Intelligence for the Interpretation of Bone Standard X-rays Prescribed by the Emergency Department (IMMEDIAT Urgences)
Acronym: IMMEDIAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 21OLE
Record Dates: First submitted 2023-04-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: Bone Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Organizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Organization (No Intervention): X-rays are done in the radiology department and the images are made available to emergency physicians without waiting for the radiologist's report, which is usually done on a delayed basis.
- Organization with AI (Other): X-rays are done in the radiology department and the images are made available to emergency physicians with the AI interpretation. X-rays flagged by IA as anormal or suspicious will be reviewed without delay by the radiologist, non-flagged X-rays will be reviewed by radiologists on a delayed basis.
  Interventions: Other: Organization with AI

INTERVENTIONS:
Other: Organization with AI — X-rays are done in the radiology department and the images are made available to emergency physicians with the AI interpretation. X-rays flagged by IA as anormal or suspicious will be reviewed without delay by the radiologist, non-flagged X-rays will be reviewed by radiologists on a delayed basis.
  Arms: Organization with AI

SUMMARY:
The study evaluates, in 3 emergency departments (ED) and on randomized alternate periods, the use of SmartUrgences®, Augmented Intelligence (AI) software to help the interpretation of bone standard X-rays prescibed by the ED.

DETAILED DESCRIPTION:
"The study evaluates, in 3 emergency departments (ED) and on randomized alternate periods, the use of SmartUrgences®, Augmented Intelligence (AI) software to help the interpretation of bone radiographs prescibed by the ED.

The primary objective of the organizational study is to evaluate, compared to the current organization for the interpretation of standard bone radiographs requested by the ED, the impact of an organization incorporating the Milvue solution, on the reduction of the patient diagnostic error rate.

A cost-consequence study is carried out, comparing from the point of view of the community (production costs according to the HAS recommendations), the radiological diagnosis within the framework of an organization with the Milvue solution, to that within the framework of the current organization without the use of the Milvue solution.

The economic study will follow the scheme of the organizational study, comparing the periods with and without the Milvue solution and analyzing the costs and consequences, by period and by patient.

This is an open-label randomized cluster multiple period cross-over study with 6 alternate periods (3 with AI, 3 with usual organization) of 1 month in each ED. The choice of the intervention for the first period will be randomized."

ELIGIBILITY:
Inclusion Criteria:

1. All adult referred by the ED for a conventional X-rays of all or part of the appendicular skeleton and/or pelvis and/or costal gril
2. Not opposed to participate"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8400 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic error rate | Through patient's discharge from the emergency department, an average of 1 day
  A diagnostic error is defined as a final consensus diagnosis that differs from the diagnosis documented in the medical record by the emergency physician prior to patient's discharge from the ED.
  A diagnostic error is defined as a final consensus diagnosis that differs from the diagnosis documented in the medical record by the emergency physician prior to patient's discharge from the ED.

SECONDARY OUTCOMES:
Time between x-ray and first diagnostic | Through patient's discharge from the emergency department, an average of 1 day
  Time between x-ray and first diagnostic, either by the emergency physician or by the radiologist
Time between x-ray and first diagnostic by the emergency physician | Through patient's discharge from the emergency department, an average of 1 day
  Time between x-ray and first diagnostic by the emergency physician in the patient medical file
Time between x-ray and final diagnostic by the emergency physician | 30 days
  Time between x-ray and final diagnostic by the emergency physician in the patient medical file. A diagnostic will be considered as final if the same as the consensus one
Rate of X-rays interpretation by radiologist without delay | 1 hour
  Rate of X-rays interpretation by radiologist without delay (i.e within 1 hour)
Number of all radiological exam per patient prescribed by the ED | Through patient's discharge from the emergency department, an average of 1 day
  Number of all radiological exam per patient prescribed by the ED (MRI, scanner, x-rays, echography)
Number of X-rays with a report by a radiologist at 30 days | 30 days
  Number of X-rays with a report by a radiologist at 30 days
Time spent in the ED by the patient | Through patient's discharge from the emergency department, an average of 1 day
  Time spent in the ED by the patient
Number of patients invited to come back in the ED | 30 days
  Number of patients invited to come back in the ED
30 days morbidity | 30 days
  New ED visit, hospitalization, radiological exam or outpatient visit, for the same reason as the first ED visit
Total cost from the hospital viewpoint | 30 days
  Total cost from the hospital viewpoint

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Saint Antoine, Paris
  - Hôpital Salpétrière, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No